CLINICAL TRIAL: NCT05295992
Title: Daily Online Adaptive Radiation Therapy of Bladder Cancer for Reduction of Intestinal Toxicity: A Prospective Trial Using an Individualized Approach and Conventional Fractionation (ARTIA-Vesica)
Brief Title: Conventionally Fractionated Adaptive Radiation Therapy of Bladder Cancer an Individualized Approach
Acronym: ARTIA-Vesica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAR-2021-06
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Muscle-Invasive Bladder Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daily Adaptive External Beam Radiation Therapy (Experimental): Daily adaptive radiation therapy delivered with Varian Ethos treatment system.
  Interventions: Device: Varian Ethos Adaptive Radiation Therapy

INTERVENTIONS:
Device: Varian Ethos Adaptive Radiation Therapy — Daily adaptive external beam radiation therapy delivered on Varian Ethos treatment system.

SUMMARY:
This is a single-arm, prospective, Phase II, multi-center clinical trial designed to demonstrate that adaptive radiotherapy for muscle invasive bladder cancer will translate into a decreased rate of acute gastrointestinal toxicity compared with the historically reported rate for non-adaptive intensity modulated radiation therapy (IMRT).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven bladder cancer
2. Urothelial carcinoma
3. Age ≥ 18 years
4. Stage T1b-T4AN0M0
5. TUR-B and PET-CT or CT of thorax/abdomen/pelvis within 8 weeks prior to inclusion
6. Suitable for radiotherapy
7. ECOG/WHO performance status 0-2
8. Written informed consent
9. For Cohort B, participant's must have normal organ and marrow function as defined below:

   * leukocytes ≥2,500/mcL
   * absolute neutrophil count ≥1,500/mcL
   * platelets ≥100,000/mcL
   * hemoglobin ≥9 g/dL
   * total bilirubin ≤ 1,5 ULN
   * AST(SGOT)/ALT(SGPT) ≤3 × ULN
   * alkaline phosphatase ≤2.5 × ULN
   * creatinine clearance <25 ml/min We recommend avoiding cisplatin for participants with creatinine clearance <50 ml/min.
   * INR and aPTT £1.5 ULN

Exclusion Criteria:

1. Prior pelvic radiation therapy
2. Inability to comply with the protocol
3. Presence of a hip prothesis
4. Grade 2 or greater baseline diarrhea
5. Uncontrolled inflammatory bowel disease (ulcerative colitis or Crohn's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Early Rate CTCAE GI Toxicity | Start of radiotherapy to 3 months after end of radiotherapy
  Change of the peak early rate of external beam radiation therapy treatment-related (CTCAE) grade 2+ diarrhea

SECONDARY OUTCOMES:
All Early CTCAE Treatment Related Toxicities | From start of radiotherapy through 3 months after end of radiotherapy
  All early adaptive radiation therapy treatment related CTCAE grade 2 and above toxicity
All Late CTCAE Treatment Related Toxicities | From 3 months after end of radiotherapy through 2 years follow-up
  All late CTCAE adaptive radiation therapy treatment related toxicity grade 2 and above
Patient Reported Outcomes (PRO) | Baseline through 2 year follow-up
  Collection of NCI PRO-CTCAE questionnaire
EORTC Quality of Life Assessment | Baseline through 2 year follow-up
  Collection of EORTC QLQ C30
EuroQol Quality of Life Assessment | Baseline through 2 year follow-up
  Collection EQ-5D-5L questionnaires
Local Progression Free Survival | From time of inclusion to local progression, assessed up to 24 months post treatment
  Local progression free survival
Local Control | At 12 and 24 months
  Local control (freedom from local progression)
Progression Free Survival | From time of inclusion to disease progression, assessed up to 24 months post treatment
  Progression free survival (from time of inclusion to disease progression)
Overall Survival | From time of inclusion to death from any cause, assessed up to 24 months post treatment
  Overall survival
Disease Free Survival | From time of inclusion to death from bladder cancer, assessed up to 24 months post treatment
  Disease Free Survival
Treatment Related Hospitalization | From of start of radiation therapy through 2 year follow-up
  Hospitalization due to adaptive radiation therapy treatment related toxicity
Workflow Feasibility | From start of radiation therapy through end of external beam treatment (approximately 6 weeks)
  Record percentage of fractions delivered with adaptive radiation therapy vs traditional IGRT

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Storm, MD, Principal Investigator — Herlev Hospital, Copenhagen University
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark